CLINICAL TRIAL: NCT05491265
Title: Impact of Intermittent Kangaroo Mother Care Versus Conventional Care Method on Vital Signs and Arterial Oxygen Saturation in Preterm Hospitalized in Neonatal Intensive Care Unit : A Randomized Controlled Trail
Brief Title: Impact of Intermittent Kangaroo Mother Care Versus Conventional Care Method on Vital Sign and Arterial Oxygen Saturation in Preterm Hospitalized in Neonatal Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Maimoona Saeed, MD Resident, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F.1-1/2015/ERB/SZABMU/955
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Kangaroo Mother Care Method
Keywords: vital signs; Intensive care

STUDY DESIGN:
Intervention Model Description: - To study the vital sign ,oxygen arterial saturation of preterm babies provided skin to skin contact versus conventional care from birth to discharge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo mother care (Experimental): To see the impact of intermittent kangaroo mother care on temperature ,oxygen saturation and heart rate.
  Interventions: Behavioral: Intermittent Kangaroo mother care
- standard of care (No Intervention): To observe temperature ,oxygen saturation and heart rate in preterm neonates not given kangaroo care

INTERVENTIONS:
Behavioral: Intermittent Kangaroo mother care — Skin to skin contact between mother and preterm newborn between gestational age 28 weeks to 36+6 weeks for three sessions per day ,each contact session of two hours .
  Arms: Kangaroo mother care

SUMMARY:
- To study the vital sign ,oxygen arterial saturation of preterm babies provided skin to skin contact versus conventional care from birth to discharge

DETAILED DESCRIPTION:
The mother and baby will be supported by a nurse and researcher. Hence, the study group mothers will be trained properly, and the required information and explanations along with displaying the video description about the KMC method will be provided for them, and the KMC will apply to their newborns.

Thus, the naked newborn, only wearing diaper and cap, was placed in a straight state between the mother's breasts and supported by a cloth bag. The caring is performed for 3 consecutive days, three times a day and each time for 2-h.

The procedure will be conducted for all samples by the head nurse and with the researcher's presence and monitoring in the morning shift, and the mothers should be supported and encouraged during the caring process. The changes in pulse ,respiration, temperature, and arterial oxygen saturation rate of the study group is controlled and recorded during the care process, at 60 min after starting the procedure and at the end of caring process before returning the newborn to the incubator. The mentioned items in the control group (conventional incubator care) should also measure and recorded simultaneously with the study group. The pulse oximetry in NICU used to measure the arterial oxygen saturation rate, and a mercury thermometer was used to measure the temperature with an auxiliary approach for 3 min. To maintain the reliability of the instrument during the research, the same pulse oximetry device and monitoring system will be applied to newborns in the same situation. The pulse oximetry probe will be taped to the toe of the left foot of all newborns

ELIGIBILITY:
Inclusion Criteria:

Birth weight between 1200 to 1800 gram Gestational age 28 weeks to 36+6 weeks Clinically stable Off oxygen support Hemodynamically stable baby No surgery performed on baby No cardiac ,nervous system problems

-

Exclusion Criteria:

Extreme preterm<28 weeks Hemodynamically unstable Underlying cardiac problems Surgical problems Those who do not give consent Unwell or hospitalized mother who is bed bound problems Gestational age 37 weeks or >37 weeks

-

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-12-03 (Estimated); Study Completion 2022-12-03 (Estimated)

PRIMARY OUTCOMES:
Temperature | 2 hours
  To measure temperature difference in babies provided with kangaroo mother care vs incubator care
Heart rate | 2 hours
  To measure heart rate variations in babies provided with kangaroo mother care vs incubator care
Oxygen Saturation | 2 hours
  To measure oxygen saturation in babies provided with kangaroo mother care vs

CONTACTS AND LOCATIONS:
Overall Officials: Dr Maimoona Saeed, MBBS, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University; Dr Fibhaa Syed, MBBS,FCPS, Study Chair — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Pakistan institute of medical sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No